CLINICAL TRIAL: NCT06448364
Title: FIRST-IN-HUMAN (FIH), OPEN-LABEL, PHASE 1 DOSE ESCALATION AND EXPANSION STUDY DESIGNED TO EVALUATE THE SAFETY, TOLERABILITY, PK, PD, AND PRELIMINARY CLINICAL ACTIVITY OF PF-07329640 AS A SINGLE AGENT OR IN COMBINATION TREATMENT FOR PARTICIPANTS WITH ADVANCED SOLID TUMORS.
Brief Title: A Study in Advanced/Metastatic Solid Tumors With the Study Medicine (PF-07329640) When Given Alone or In Combination
Acronym: LTbR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic business decision
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5181001
Record Dates: First submitted 2024-04-17; First posted 2024-06-07 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Advanced or Metastatic Solid Tumors; Non-Small Cell Lung Cancer; Colorectal Cancer; Urothelial Cancer; Melanoma
Keywords: Solid tumors; metastatic; advanced; micro satellite stable; anti-VEG; anti-PD-1; PF-07329640; LTbetaR; LTbR; sasanlimab; bevacizumab; PD-1 resistance; PD-1 naive; PDx resistance; PDxnaive; Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal; Non-Muscle Invasive Bladder Cancer (NMIBC); Non-Muscle-Invasive Bladder Cancer; Malignant Melanoma; Microsatellite Stable Colorectal Cancer (MSS CRC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Melanoma; Neoplasm Metastasis; Non-Muscle Invasive Bladder Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1A: PF-07329640 (αLTβR) Monotherapy (Experimental): PF-07329640 (αLTβR) monotherapy at prescribed dose and frequency in 28-day cycles
  Interventions: Biological: PF-07329640
- Part 1B: PF-07329640 (αLTβR) + bevacizumab (Experimental): PF-07329640 (αLTβR) + bevacizumab dose escalation in NSCLC and MSS CRC at prescribed dose and frequency in 28-day cycles
  Interventions: Biological: PF-07329640; Biological: bevacizumab
- Part 1C: PF-07329640 (αLTβR) + sasanlimab (Experimental): PF-07329640 (αLTβR) + sasanlimab dose escalation in NSCLC, melanoma, UC, and MSS CRC at prescribed dose and frequency in 28-day cycles
  Interventions: Biological: PF-07329640; Biological: sasanlimab
- Part 2A: PF-07329640 (αLTβR) + bevacizumab (Experimental): PF-07329640 (αLTβR) + bevacizumab dose expansion in NSCLC 2L+ and MSS CRC 2L+ at prescribed dose and frequency in 28-day cycles
  Interventions: Biological: PF-07329640; Biological: bevacizumab
- Part 2B: PF-07329640 (αLTβR) + sasanlimab (Experimental): PF-07329640 (αLTβR) + sasanlimab dose expansion in NSCLC, melanoma, UC, and MSS CRC at prescribed dose and frequency in 28-day cycles
  Interventions: Biological: PF-07329640; Biological: sasanlimab
- Part 2C: PF-07329640 (αLTβR) + SOC (Experimental): PF-07329640 (αLTβR) + SOC (anti-PD-1+ platinum-based chemo) dose expansion for αPDx-naïve NSCLC 1L at prescribed dose and frequency in 28-day cycles
  Interventions: Biological: PF-07329640
- Part 2D: PF-07329640 (αLTβR) (Experimental): PF-07329640 (αLTβR) dose expansion in advanced solid tumors at prescribed dose and frequency in 28-day cycles
  Interventions: Biological: PF-07329640

INTERVENTIONS:
Biological: PF-07329640 — an anti-lymphotoxin beta receptor agonist
  Other Names: LtbR, LTbetaR
Biological: sasanlimab — A monoclonal antibody that blocks the interaction between PD-1 and PD-L1/L2
  Other Names: PF-06801591
  Arms: Part 1C: PF-07329640 (αLTβR) + sasanlimab; Part 2B: PF-07329640 (αLTβR) + sasanlimab
Biological: bevacizumab — a monoclonal antibody that blocks VEGF
  Other Names: Zirabev; Bevacizumab-bvzr
  Arms: Part 1B: PF-07329640 (αLTβR) + bevacizumab; Part 2A: PF-07329640 (αLTβR) + bevacizumab

SUMMARY:
The purpose of this study is to learn about the safety (the impact of the study drug on the participant's body), effects of the study drug alone or in combination with bevacizumab or sasanlimab, and to find the best dose.

This study is seeking participants who have solid tumors that:

* have advanced (cancer that doesn't disappear or stay away with treatment) or
* has spread to other parts of the body (metastatic).

This includes (but limited to) the following cancer types:

* Non-Small Cell Lung Cancer (NSCLC): It's a type of lung cancer where the cells grow slowly but often spread to other parts of the body.
* Colorectal Cancer (CRC): This is a disease where cells in the colon or rectum grow out of control.
* Urothelial Cancer (UC): This is a cancer that starts in the urinary systems.
* Melanoma: Skin cancer that develops when melanocytes (the cells that give the skin its tan or brown color) start to grow out of control.

All participants in this study will receive the study medication (PF-07329640) as an IV infusion (given directly into a vein) at the study clinic every week for repeating 28-day cycles.

Depending on which part of the study participants are enrolled in they will receive the study medication (PF-07329640 alone or in combination with other anti-cancer medications (bevacizumab or sasanlimab). Bevacizumab is given in the clinic as IV infusion every two weeks and sasanlimab is given as a shot under the skin every 4 weeks.

Participants can continue to take the study medication (PF-07329640) and bevacizumab until their cancer is no longer responding. Participants who are taking sasanlimab may receive it for up to 2 years.

The study will look at the experiences of people receiving the study medicines. This will help see if the study medicines are safe and effective.

Participants will be involved in this study for up to 4 years. During this time, they will have a study visit every week. After they have stopped taking the study medication (at about at 2 years) they will be followed for another two years to see how they are doing.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced, unresectable, and/or metastatic or relapsed/refractory solid tumor
* Part 1:

  * Part 1A: Participants with solid tumors where anti-PD-(L)1 is an established treatment. Participants must have progressed on or following prior anti-PD-(L)1 therapy if approved, available, tolerable, and eligible.
  * Part 1B & C: Participants either meeting Part 1A criterion, or participants with "cold" solid tumors where anti-PD-(L)1 therapy is not an established treatment
* Part 2:

  * Part 2A:
  * Cohort 1: Participants with NSCLC must have received platinum-based chemotherapy and anti-PD-(L)1 or have intolerability to or refusal of standard therapies. NSCLC participants with known activating mutation(s) must also have received prior approved and available targeted therapy(ies) for the associated mutation(s) or have intolerability or documented refusal of these therapies.
  * Cohort 2: Participants with MSS CRC must have received at least fluoropyrimidine-, oxaliplatin, and irinotecan-based chemotherapy, an anti-VEGF agent (if not receiving anti-VEGF on protocol), and anti-epidermal growth factor receptor (EGFR) inhibitor (if RAS wildtype) and/or other molecularly targeted therapy if appropriate.
  * Part 2B:

    * NSCLC (2L+) participants as described above in Part 2A
    * MSS CRC (2L+) participants as described above in Part 2A
    * UC (2L+) participants must have received prior platinum-based chemotherapy, anti-PD-(L)1 therapy, or enfortumab vedotin.
  * Part 2C; anti-PDx naive NSCLC (1L) participants must not have received standard of care therapy with anti-PD-(L)1.
* At least 1 measurable lesion based on RECIST 1.1 that has not been previously irradiated (Part 1 exceptions permitted after review and approval)
* Able to provide pre-treatment (and optional on-treatment) tumor tissue
* Resolution of acute effects of any prior therapy to either baseline or CTCAE Grade 1

Exclusion Criteria:

* Treatment with any systemic anticancer therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to planned first dose
* Prior treatment with another anti-LTβR agonist
* Systemic anticancer therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to planned first dose (6 weeks for mitomycin C or nitrosoureas). Prior targeted or endocrine therapy require an interval of 2 weeks or 5 half-lives (whichever is shorter) prior to planned first dose.
* Lack of adequate organ (bone marrow, renal, liver) function
* Active infection requiring systemic treatment.
* Active or history of autoimmune disease (eg, systemic lupus erythematosus, rheumatoid arthritis) requiring chronic systemic steroid or immune-modulatory therapy (not including oral physiological replacements)
* History of Grade ≥3 immune mediated adverse event (AE) (including aspartate aminotransferase (AST)/alanine aminotransferase (ALT) elevations that were considered drug related) and/or CRS that was considered related to prior immune-modulatory therapy and required immunosuppressive therapy.
* Known or suspected hypersensitivity to any PF-07329640 components, or to monoclonal antibodies (mAbs) or other therapeutic proteins such as fresh frozen plasma, human serum albumin, cytokines, or interleukin, or anti-PD-(L)1 therapy (the latter applicable for Part 1C and Part 2B/C participants only
* Brain metastasis or primary brain tumor requiring immediate local intervention (surgery, radiosurgery) in the opinion of the investigator.
* Other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix, Bowen's disease. Presence of other indolent cancer requires prior sponsor approval.
* Organ transplant requiring immunosuppressive treatment or prior allogeneic bone marrow or hematopoietic stem cell transplant.
* Pregnant or breastfeeding
* Persistent or recurring ≥ Grade 2 neuropathy prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
PART 1: Number of participants with Dose-limiting toxicities (DLT) | First cycle, Day 1 up to Day 28
  Any of the prespecified AEs that are attributable to one, the other, or both study treatments, occurring in the DLT observation period are considered DLTs, excluding toxicities clearly due to underlying disease or extraneous causes:
PART 1 & 2: Incidence of Adverse Events (AE)s | From start of the treatment up to 90 days after last dose or start of new anticancer therapy, whichever occurred first
  An adverse event (AE) was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/ incapacity; congenital anomaly. AEs included both serious and all non-serious AEs.
To: PART 1 & 2: Number of participants with laboratory abnormalities | From start of treatment up to 90 days after last dose or start of new anticancer therapy, whichever occurred first
  Number of participants with laboratory test abnormalities. Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes, clinical chemistry, and urinalysis (dipstick and microscopy).
Part 2: "Objective Response - Number of Participants With Objective Response " | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion, approximately 2 years'
  Percentage of participants with objective response-based best overall response (BOR) of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by the Investigator.

SECONDARY OUTCOMES:
Part 1: Objective Response - Number of Participants With Objective Response | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion, approximately 2 years
  Percentage of participants with objective response-based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by the Investigator
Time to event endpoints: duration of response (DOR) by RECIST v1.1 | Baseline to confirmed disease progression, up to 2 years after the last dose of study treatmennt
  Time to event: DOR according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as assessed by the Investigator.
Time to event endpoints: progression-free survival (PFS) by RECIST v1.1 | Baseline to confirmed disease progression, up to 2 years after the last dose of study treatmennt
  Time to event: PFS according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as assessed by the Investigator.
Part 1A: Maximum Observed Serum Concentration (Cmax) of PF-07329640 | Cycle 1 Day 1 & Cycle 2 Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, End of Infusion (EOI), 4, and 8 hours Cycle 2: Pre-dose, EOI, 4, and 8 hours
Part 1A: Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-07329640 | Cycle 1 Day 1 & Cycle 2 Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, End of Infusion (EOI), 4, and 8 hours Cycle 2: Pre-dose, EOI, 4, and 8 hours
Part 1A: Serum Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-07329640 | Cycle 1 Day 1 & Cycle 2 Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, End of Infusion (EOI), 4, 8, 24, 48, 72 hours post-dose (Day 1-4); Pre-dose, EOI, 4 hours post-dose (Day 8); pre-dose, EOI (Day 15) Cycle 2: Pre-dose, EOI, 4, 8, 24, 48, 72 hours post-dose (Day 1-4); Pre-dose, and 4 hours post-dose (Day 15)
Serum Concentrations of PF-07329640 in combination (Part 1B/1C/2A/2B/2C) | pre-dose and end of infusion on Cycle 1 Day 1, Cycle 1Day 15, Cycle 2 Day 1 (Each cycle is 28 days)
  comparison Predose and end of infusion blood serum concentrations at Cycle 1 day 1 and 15, and Cycle Day 1
Incidence and titers of antidrug antibodies (ADA) against PF-07329640 | Baseline though study completion, an average of 2 years
  the number of patients with ADAs against PF-07329640 and the concentration of those ADAs
Paired Tumor Biopsies | Baseline through Cycle 2 Day 15 (each cycle is 28 days)
  Changes in quantity and maturation state of tertiary lymphoid structure (TLS)s in tumor biopsy tissues at Cycle 2 Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (4):
  - Highlands Oncology, Fayetteville, Arkansas
  - Highlands Oncology, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - NEXT Oncology, San Antonio, Texas
- Puerto Rico (3):
  - Hospital Oncológico Dr. Isaac González-Martinez, Rio Piedras
  - Pan American Center for Oncology Trials, LLC, Rio Piedras
  - Pan American Center for Oncology Trials- Hospital Oncologico, Rio Piedras

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5181001